CLINICAL TRIAL: NCT03515811
Title: To Confirm the Safety and Performance of the Signia™ Stapling System Using Signia™ Intelligent Loading Units With Tri-Staple™ 2.0 Intelligent Reloads in Abdominal and Thoracic Procedures.
Brief Title: A Post Market Study to Confirm the Safety and Performance of the Signia™ Stapling System.
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT17025SIG
Record Dates: First submitted 2018-04-23; First posted 2018-05-04 (Actual); Results first posted 2023-03-31 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Abdominal Injury; Thoracic Diseases
MeSH Terms: conditions — Abdominal Injuries; Thoracic Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Abdominal: Signia™ Stapling System using Signia™ Intelligent Loading Units with Tri-Staple™ 2.0 Intelligent Reloads.
  Abdominal (approximately 53 subjects).
  Interventions: Device: Signia™ Stapling System
- Thoracic: Signia™ Stapling System using Signia™ Intelligent Loading Units with Tri-Staple™ 2.0 Intelligent Reloads.
  Thoracic (approximately 74 subjects).
  Interventions: Device: Signia™ Stapling System

INTERVENTIONS:
Device: Signia™ Stapling System — Signia™ Stapling System using Signia™ Intelligent Loading Units with Tri- Staple™ 2.0 Intelligent Reloads.

SUMMARY:
The objectives of this prospective, two-arm, multicenter post-market study is to confirm safety and performance through the incidence of subjects reporting serious adverse device effects (ADEs) up to and including 30 days following use of Signia™ Stapling System with Endo GIA™ with Tri-Staple™ Technology and Tri-Staple™ 2.0 Intelligent Reloads in subjects undergoing indicated abdominal or thoracic procedures for resection, transection and creation of anastomosis per the IFU.

DETAILED DESCRIPTION:
This study will evaluate the use of Signia™ Stapling System using Signia™ Intelligent Loading Units with Tri-Staple™ 2.0 Intelligent Reloads in indicated abdominal or thoracic procedures (e.g., resection, transection of tissue, and creation of anastomoses). Subjects who meet the eligibility criteria will be considered for study participation at a minimum of 10 sites and will be followed up to and including 30 days post-operative. Overall the study is estimated to progress for up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (male or female) between 22 and 80 years of age inclusive at the time of the procedure.
2. The subject must be willing and able to participate in the study procedures and to understand and sign the informed consent.
3. The subject is scheduled to undergo an indicated primary abdominal or thoracic procedure for resection, transection and creation of anastomosis per the IFU where the Signia™ Stapling System with Endo GIA™ with Tri-Staple™ Technology and Tri-Staple™ 2.0 Intelligent Reloads will be used per its IFU.Additionally, if considered appropriate for the procedure only Medtronic buttresses can be used during the course of the study.

3a. Thoracic procedures may include, but are not limited to wedge resection and lobectomy, and may include video assisted thoracic surgery (VATS) or open procedures.

3b. Abdominal procedures may include, but are not limited to, laparoscopic sleeve gastrectomy (LSG), laparoscopic Roux-en-Y gastric bypass (LRYGB).

Exclusion Criteria:

1. Subjects undergoing cardiac and vascular procedures.
2. The procedure is an emergency procedure.
3. The procedure is a revision/reoperation of a primary operation..
4. Any female subject who is pregnant. 4a. Females of child-bearing potential will be required to undergo either a urine pregnancy test or serum pregnancy test during Screening and confirmed on the day of operation (except for subjects who are surgically sterile or are post-menopausal for at least two years) (USA only) and per EU local requirements.
5. Any subject who is considered to be part of a vulnerable population (e.g. prisoners or those without sufficient mental capacity).
6. The subject is unable or unwilling to comply with the study requirements or follow-up schedule.
7. The subject has comorbidities which, in the clinical judgment of the Investigator, will not be appropriate for the study or the subject has an estimated life expectancy of less than 6 months.
8. The subject has been diagnosed with a bleeding disorder and/or is undergoing active and not reversed anticoagulant treatment.
9. The subject is concurrently enrolled in another investigational drug or device research study or has been enrolled in another study within 30 days of enrollment.
10. Pre-existing/chronic conditions specific to Tri-Staple™ 2.0 Reload contraindications as described in the IFU.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 74 Thoracic subjects arm 53 abdominal subjects arm
Sampling Method: Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2020-07-13 (Actual); Study Completion 2020-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelley Kennedy, Study Director — Medtronic
Locations (11):
- United States (6):
  - Cedars Sinai Medical Center, Los Angeles, California
  - Albany Medical College, Albany, New York
  - WakeMed Bariatric Specialists of North Carolina, Cary, North Carolina
  - UNC Chapel Hill, Chapel Hill, North Carolina
  - Duke Regional Hospital, Durham, North Carolina
  - Inova Fairfax Hospital, Falls Church, Virginia
- Institut Universitaire de Cardiologie et de Pneumologie de Quebec, Québec, Quebec, Canada
- Azienda Ospedaleria San Gerardo, Monza, Italy
- Spain (2):
  - Hospital Universitario del Rocio, Seville
  - Hospital Universitario Virgen Macarena, Seville
- Blackpool Victoria Hospital, Blackpool, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Abdominal: Signia™ Stapling System using Signia™ Intelligent Loading Units with Tri-Staple™ 2.0 Intelligent Reloads.
  Abdominal (approximately 53 subjects).
  Signia™ Stapling System: Signia™ Stapling System using Signia™ Intelligent Loading Units with Tri- Staple™ 2.0 Intelligent Reloads.
- Thoracic: Signia™ Stapling System using Signia™ Intelligent Loading Units with Tri-Staple™ 2.0 Intelligent Reloads.
  Thoracic (approximately 74 subjects).
  Signia™ Stapling System: Signia™ Stapling System using Signia™ Intelligent Loading Units with Tri- Staple™ 2.0 Intelligent Reloads.
Period: Overall Study
Arm/Group | Abdominal | Thoracic
Started | 51 | 85
Completed | 46 | 77
Not Completed | 5 | 8
Not completed — Lost to Follow-up | 2 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Death | 1 | 1
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Technical Problems | 1 | 0
Not completed — Subject Unable to Return for Follow-Up | 0 | 2
Not completed — COVID-19 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Abdominal | Thoracic | Total
Number analyzed (Participants) | 51 | 85 | 136
Age, Continuous [Median (Standard Deviation); unit: years] | 48.0 (13.25) | 68.0 (10.16) | 62.5 (14.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 35 | 75
  Male | 11 | 50 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 5 | 19
  Not Hispanic or Latino | 37 | 49 | 86
  Unknown or Not Reported | 0 | 31 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 4 | 15
  White | 38 | 79 | 117
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 0 | 5 | 5
  United States | 38 | 38 | 76
  Italy | 0 | 18 | 18
  United Kingdom | 0 | 13 | 13
  Spain | 13 | 11 | 24
Pregnancy Test Performed [Count of Participants; unit: Participants] — Population: Pregnancy test was only performed for female subjects of child-bearing age and potential.
  Participants
    number analyzed (Participants) | 40 | 35 | 75
    (all) | 20 | 7 | 27

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint is the Number of Subjects Reporting Serious Adverse Device Effects (SADEs), Including Intra- and Post-operative Leaks.
Description: The primary endpoint is the number of subjects reporting serious adverse device effects (SADEs) up to and including 30 days, including intra- and post-operative leaks. A Serious Adverse Device Effect (SADE) is an adverse event related to the use of an investigational medical device, that is deemed serious in nature. To be deemed serious, and adverse event must meet one or more of the following criteria:
  Led to a death, b. Led to a serious deterioration in the health of the subject, that either resulted in:
  1. Resulted in a life-threatening illness or injury, or
  2. Resulted in a permanent impairment of a body structure or a body function, or
  3. In-patient or prolonged hospitalization, or
  4. Medical or surgical intervention to prevent life threatening illness or injury or permanent impairment to a body structure or a body function, or c. Led to fetal distress, fetal death or a congenital abnormality or birth defect.
Time Frame: Up to and including 30 days intra- and post-operative.
Measure: Count of Participants; unit: Participants
Groups:
- Abdominal: Signia™ Stapling System using Signia™ Intelligent Loading Units with Tri-Staple™ 2.0 Intelligent Reloads.
  Abdominal (approximately 53 subjects).
  Signia™ Stapling System: Signia™ Stapling System using Signia™ Intelligent Loading Units with Tri- Staple™ 2.0 Intelligent Reloads.
  95% Confidence Interval: (0.0%-7.0%)
- Thoracic: Signia™ Stapling System using Signia™ Intelligent Loading Units with Tri-Staple™ 2.0 Intelligent Reloads.
  Thoracic (approximately 74 subjects).
  Signia™ Stapling System: Signia™ Stapling System using Signia™ Intelligent Loading Units with Tri- Staple™ 2.0 Intelligent Reloads.
  95% Confidence Interval: (5.0%-19.2%).
Arm/Group | Abdominal | Thoracic
Number analyzed (Participants) | 51 | 85
Participants | 0 | 9
Statistical Analysis 1: Comparison: Thoracic; Test type: Other; Percentage and confidence interval = 10.6, 95% CI 2-sided [5.0 to 19.2] — 95% CI: 5.0%-19.2%
Statistical Analysis 2: Comparison: Abdominal; Test type: Other; Percentage and confidence interval = 0.0, 95% CI 2-sided [0.0 to 7.0] — 95% CI: 0.0%-7.0%

2. Primary Outcome: The Primary Endpoint is the Number of Subjects Reporting Serious Adverse Device Effects (SADEs), Including Intra- and Post-operative Leaks.
Description: The primary endpoint is the number of subjects reporting serious adverse device effects (SADEs), including intra- and post-operative leaks up to and including 30 (+14) days post-procedure. A Serious Adverse Device Effect (SADE) is an adverse event related to the use of an investigational medical device, that is deemed serious in nature. To be deemed serious, and adverse event must meet one or more of the following criteria:
  Led to a death, b. Led to a serious deterioration in the health of the subject, that either resulted in:
  1. Resulted in a life-threatening illness or injury, or
  2. Resulted in a permanent impairment of a body structure or a body function, or
  3. In-patient or prolonged hospitalization, or
  4. Medical or surgical intervention to prevent life threatening illness or injury or permanent impairment to a body structure or a body function, or c. Led to fetal distress, fetal death or a congenital abnormality or birth defect.
Time Frame: Up to and including 30 (+14) days post-procedure.
Measure: Count of Participants; unit: Participants
Groups:
- Overall: Overall subjects included in the study, in both the thoracic and abdominal indications.
Arm/Group | Overall
Number analyzed (Participants) | 136
Participants | 9
Statistical Analysis 1: Comparison: Overall; Test type: Other; Percentage and confidence interval = 6.6, 95% CI 2-sided [3.1 to 12.2] — 95% CI: 3.1%-12.2%

3. Secondary Outcome: The Secondary Endpoint is Device Deficiencies/Malfunctions Affecting the Intended Performance of the Device.
Description: The secondary endpoint is device deficiencies/malfunctions affecting the intended performance of the device. All recorded device deficiencies/malfunctions were captured and assessed by the Investigator. A Device Deficiency is defined as inadequacy of a medical device with respect to its identity, quality, durability, reliability, safety or performance.
  Note: Device deficiencies include malfunctions, use errors, and inadequate labeling.
Time Frame: Up to and including 30 (+14) days post-operative.
Measure: Count of Participants; unit: Participants
Arm/Group | Abdominal | Thoracic
Number analyzed (Participants) | 51 | 85
Participants | 2 | 2

4. Secondary Outcome: The Secondary Endpoint is the Intra-operative Staple Line Assessment Assessing: Staple Line Integrity (B Formation).
Description: The secondary endpoint is device deficiency/malfunctions affecting the intended performance of the device including: intra- and post-operative staple line assessments. B formation is defined as consistent formation of the staple-line fired by the Signia Stapling System handle.
Time Frame: Up to and including 30 (+14) days post-operative.
Population: 36 subjects had intra-operative assessment data incorrectly recorded for B-formation, so this data was excluded from this part of the intra-operative analysis results. Thus, the overall number of participants analyzed is different for this parameter (44 for abdominal, and 56 for thoracic).
Measure: Count of Participants; unit: Participants
Arm/Group | Abdominal | Thoracic
Number analyzed (Participants) | 44 | 56
Participants | 44 | 55

5. Secondary Outcome: The Secondary Endpoint is the Intra-operative Staple Line Assessment Assessing: Number of Staple-line Bleeding (Measured as > 50 cc) Occurrences.
Description: The secondary endpoint is device deficiency/malfunctions affecting the intended performance of the device including: intra- and post-operative staple line assessments. Number of staple-line bleeding (measured as > 50 cc) refers to occurrences of bleeding at the staple-line only, and not in the study procedure as a whole.
Time Frame: Up to and including 30 (+14) days post-operative.
Population: One abdominal subject died during their study procedure, so the Overall Number of Participants Analyzed in the Abdominal group dropped from 51 to 50 for the intra-operative assessments, since their staple-line was not assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | Abdominal | Thoracic
Number analyzed (Participants) | 50 | 85
Participants | 0 | 0

6. Secondary Outcome: The Secondary Endpoint is the Intra-operative Staple Line Assessment Assessing: Additional Interventions to Treat Staple-line Failure.
Description: The secondary endpoint is device deficiency/malfunctions affecting the intended performance of the device including: intra- and post-operative staple line assessments. Examples of additional interventions to treat staple-line failure include: glue, manual over sew, Medtronic buttress as additional reinforcement, or intraoperative revision/recreation of the anastomosis.
Time Frame: Up to and including 30 (+14) days post-operative.
Measure: Count of Participants; unit: Participants
Arm/Group | Abdominal | Thoracic
Number analyzed (Participants) | 51 | 85
Participants | 3 | 42

7. Secondary Outcome: The Secondary Endpoint is the Intra-operative Staple Line Assessment Assessing: Number of Intra-operative Leakage.
Description: The secondary endpoint is device deficiency/malfunctions affecting the intended performance of the device including: intra- and post-operative staple line assessments. Number of intra-operative leakage as measured by air leak test performed by the surgeon, or standard of care, as applicable.
Time Frame: Up to and including 30 (+14) days post-operative.
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Abdominal | Thoracic
Number analyzed (Participants) | 50 | 85
Participants | 0 | 5

8. Secondary Outcome: The Secondary Endpoint is the Post-operative Surgical Site Assessment Assessing: Number of Post-operative Leakage.
Description: The secondary endpoint is device deficiency/malfunctions affecting the intended performance of the device including: intra- and post-operative staple line assessments. Number of post-operative leakage as evidenced confirmed by imaging, subject presentation or decline in status, or need for re-operation/re-intervention.
Time Frame: Up to and including 30 (+14) days post-operative.
Measure: Count of Participants; unit: Participants
Arm/Group | Abdominal | Thoracic
Number analyzed (Participants) | 51 | 85
Participants | 0 | 7

9. Secondary Outcome: The Secondary Endpoint is the Post-operative Surgical Site Assessment Assessing: Duration of Air Leakage >7 Days.
Description: The secondary endpoint is device deficiency/malfunctions affecting the intended performance of the device including: intra- and post-operative staple line assessments. Prolonged air leaks are considered >7 days in duration.
Time Frame: Up to and including 30 (+14) days post-operative.
Population: Duration of air leakage was not assessed in the abdominal group, becasue there were no air leaks in the abdominal group.
Measure: Count of Participants; unit: Participants
Arm/Group | Abdominal | Thoracic
Number analyzed (Participants) | 0 | 85
Participants | 0 | 3

10. Secondary Outcome: The Secondary Endpoint is the Post-operative Surgical Site Assessment Assessing: Number of Post-operative Infection.
Description: The secondary endpoint is device deficiency/malfunctions affecting the intended performance of the device including: intra- and post-operative staple line assessments. Number of post-operative infection was assessed by the Investigator according to the standard of care and site policy, ex. Positive wound culture.
Time Frame: Up to and including 30 (+14) days post-operative.
Measure: Count of Participants; unit: Participants
Arm/Group | Abdominal | Thoracic
Number analyzed (Participants) | 51 | 85
Participants | 1 | 8

11. Secondary Outcome: The Secondary Endpoint is the Post-operative Surgical Site Assessment Assessing: Additional Interventions to Treat Staple-line Failure.
Description: as for outcome 6
Time Frame: Up to and including 30 (+14) days post-operative.
Measure: Count of Participants; unit: Participants
Arm/Group | Abdominal | Thoracic
Number analyzed (Participants) | 51 | 85
Participants | 0 | 2

12. Secondary Outcome: The Secondary Endpoint is the Post-operative Surgical Site Assessment Assessing: Number of Repeat Hospital Admissions for Primary Procedure-related Complications.
Description: The secondary endpoint is device deficiency/malfunctions affecting the intended performance of the device including: intra- and post-operative staple line assessments. The number of repeat hospital admissions for primary procedure-related complications was assessed.
Time Frame: Up to and including 30 (+14) days post-operative.
Measure: Count of Participants; unit: Participants
Arm/Group | Abdominal | Thoracic
Number analyzed (Participants) | 51 | 85
Participants | 1 | 4

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to and including 30 (+14) days post-procedure.
Arm/Group | Abdominal | Thoracic
All-Cause Mortality (participants affected / at risk) | 1/51 | 1/85
Serious Adverse Events (participants affected / at risk) | 6/51 | 21/85
Other Adverse Events (participants affected / at risk) | 0/51 | 31/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abdominal (N=51) | Thoracic (N=85)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Arterial haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 3 (3)
Arterial injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bronchial injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Brain injury (Nervous system disorders) | 0 (0) | 1 (1)
Device leakage (Product Issues) | 0 (0) | 1 (1)
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 8 (8)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abdominal (N=51) | Thoracic (N=85)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 15 (15)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 (0) | 9 (9)
Post-operative leak (Surgical and medical procedures) | 0 (0) | 7 (10)

LIMITATIONS AND CAVEATS:
There were no limitations or caveats in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-08-10): https://cdn.clinicaltrials.gov/large-docs/11/NCT03515811/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-08): https://cdn.clinicaltrials.gov/large-docs/11/NCT03515811/SAP_001.pdf